CLINICAL TRIAL: NCT02384148
Title: Measure and Comparison of Molecular Circadian Clock Properties in Healthy Subjects, Obese and Type 2 Diabetic Patients.
Brief Title: Study of Circadian Clock Properties in Healthy Subjects, Obese and Type 2 Diabetic Patients.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Charna Dibner, phD, University Hospital, Geneva
Other Study IDs: 11-015
Record Dates: First submitted 2015-02-27; First posted 2015-03-10 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-12

CONDITIONS: Circadian Rhythm; Diabetes; Obesity
MeSH Terms: conditions — Diabetes Mellitus; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (4):
- Healthy: Healthy volunteers with no inflammation diseases, no neoplasia, no allergy to lidocaine.
  Interventions: Other: Circadian rhythm measurement; Procedure: Skin biopsy
- Type 2 diabetic non obese: Type 2 diabetic patients with HbA1c>6.5%, body mass index 19-30 kg/m2, no inflammation diseases, no neoplasia, no allergy to lidocaine.
  Interventions: Other: Circadian rhythm measurement; Procedure: Skin biopsy
- Type 2 diabetic obese: Type 2 diabetic patients with HbA1c>6.5%, body mass index >30 kg/m2, no inflammation diseases, no neoplasia, no allergy to lidocaine.
  Interventions: Other: Circadian rhythm measurement; Procedure: Skin biopsy
- obese: Obese non diabetic patients with HbA1c<6.5%, body mass index >30 kg/m2, no inflammation diseases, no neoplasia, no allergy to lidocaine.
  Interventions: Other: Circadian rhythm measurement; Procedure: Skin biopsy

INTERVENTIONS:
Other: Circadian rhythm measurement
Procedure: Skin biopsy — A 2mm diameter skin biopsy is performed by a physician using standard procedure.

SUMMARY:
The investigators aimed to characterize human circadian clockwork in healthy individuals in comparison to obese and type 2 diabetic subjects, employing the noninvasive experimental approach allowing the study of circadian profile in human individuals.

DETAILED DESCRIPTION:
The investigators specifically aim to obtain and analyze the circadian profile of skin fibroblasts from healthy, obese and T2D subjects. Does circadian oscillator profile and its parameters (phase, period and amplitude) will differ between healthy individuals and obese/ T2D patients? Skin biopsy will be performed in order to collect and culture skin fibroblast cells.

In vivo bioluminescence recording will be performed in primary human skin fibroblast cells. The profiles obtained from 10 subjects in each group will be compared to their healthy counterparts.

Bmal1and Per2 are clock genes. Lentiviral transduction of Bmal1-luciferase or Per2-luciferase in fibroblasts allow observation of circadian oscillations using bioluminescence assay. Phase, period length and amplitude are used to characterize the circadian rhythm.

ELIGIBILITY:
Inclusion Criteria:

* age 20-80
* consent obtained

Exclusion Criteria:

* neoplasia
* inflammatory disease
* allergy to lidocaine

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: One hundred normolipidemic healthy individuals, one hundred T2D subjects divided into two sub-groups (T2D non-obese and T2D obese) and one hundred obese non diabetic patients will be included.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2011-06; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Difference of period length | 5 days
  Period length will be calculated from oscillation profiles of Bmal1-luciferase or Per2-luc luciferase.

SECONDARY OUTCOMES:
Difference of amplitude | 5 days
  Amplitude will be calculated from oscillation profiles of Bmal1-luciferase or Per2-luc luciferase.

CONTACTS AND LOCATIONS:
Locations (1):
- Geneva University Hospital, Geneva, Switzerland

REFERENCES:
- [Background] Pagani L, Schmitt K, Meier F, Izakovic J, Roemer K, Viola A, Cajochen C, Wirz-Justice A, Brown SA, Eckert A. Serum factors in older individuals change cellular clock properties. Proc Natl Acad Sci U S A. 2011 Apr 26;108(17):7218-23. doi: 10.1073/pnas.1008882108. Epub 2011 Apr 11. PMID 21482780
- [Background] Brown SA, Fleury-Olela F, Nagoshi E, Hauser C, Juge C, Meier CA, Chicheportiche R, Dayer JM, Albrecht U, Schibler U. The period length of fibroblast circadian gene expression varies widely among human individuals. PLoS Biol. 2005 Oct;3(10):e338. doi: 10.1371/journal.pbio.0030338. Epub 2005 Sep 27. PMID 16167846